CLINICAL TRIAL: NCT02543099
Title: The Effect of Policosanol on Elderly Patients With Endothelial Dysfunction
Brief Title: Efficacy and Safety Study of Policosanol
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20150811
Record Dates: First submitted 2015-08-30; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Endothelial Dysfunction
Keywords: endothelial function; policosanol; efficacy; safety
MeSH Terms: interventions — policosanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- policosanol (Experimental): Patients will receive policosanol 20mg daily until the end of the trial.
  Interventions: Drug: policosanol
- placebo (Placebo Comparator): Patients will receive placebo 20mg daily until the end of the trial;
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: policosanol — Patients will receive policosanol 20mg Qd
  Other Names: PPG; Lipex; dupla; ateromixol
  Arms: policosanol
Drug: placebo — Patients will receive placebo 20mg Qd;
  Arms: placebo

SUMMARY:
The purpose of this study is to assess the clinical efficacy and safety of policosanol on elderly patients with endothelial dysfunction

DETAILED DESCRIPTION:
100 selected elderly patients with endothelial dysfunction were randomized to two groups,Group1:received policosanol 20mg qd;Group2:received placebo 20mg qd；endothelial function was tested by peripheral arterial tonometry(PAT) before and after 6 months' treatment with policosanol or placebo respectively; Endothelial dysfunction is defined as reactive hyperemia index(RHI)< 1.67; The aim of this study is to assess the clinical efficacy and safety of policosanol on elderly patients with endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 60 years old；
2. Patients with endothelial dysfunction
3. Provision of informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Acute myocardial infarction ,severe trauma , major operation or stroke within six months;
2. Tumor or inflammatory diseases
3. Known allergies to policosanol
4. Life expectancy less than 1 year
5. secondary dyslipidemia 6.taking other experimental medicine within six months;

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
reactive hyperemia index (RHI) measured by Endo-PAT | 6 months after the treatment with policosanol or placebo
  Novel digital pulse amplitude tonometry (PAT) offers the possibility of an easy and rapid assessment of vascular function. Endothelial function was assessed using a Endo-PAT device (Itamar Medical Ltd, Caesarea, Israel)and recorded as a reactive hyperemia index (RHI)

SECONDARY OUTCOMES:
Effects of Policosanol in Older Patients | 6 months after the treatment with policosanol or placebo
  Triglyceride(TG),total cholesterol (TC), low-density lipoprotein(LDL-C), high- density lipoprotein cholesterol (HDL-C ), lipoprotein (a), apolipoprotein AI (apo AI) and apolipoprotein B (apo B) were measured at the clinical biochemistry.
the safety of policosanol evaluated by clinical and statistical analysis, including clinical adverse reactions, laboratory indexes (such as liver function, kidney function and creatine kinase (CK) value) and vital signs | 6 months after the treatment with policosanol or placebo
  The safety was evaluated by clinical and statistical analysis, including clinical adverse reactions, laboratory indexes (such as liver function, kidney function and creatine kinase (CK) value) and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: ping ye, M.D, Principal Investigator — Department of geriatric Cardiology, Chinese PLA general hospital
Locations (1):
- Division of South, General Hospital of Chinese People's Armed Police Forces, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Reriani MK, Lerman LO, Lerman A. Endothelial function as a functional expression of cardiovascular risk factors. Biomark Med. 2010 Jun;4(3):351-60. doi: 10.2217/bmm.10.61. PMID 20550469
- [Result] Affuso F, Ruvolo A, Micillo F, Sacca L, Fazio S. Effects of a nutraceutical combination (berberine, red yeast rice and policosanols) on lipid levels and endothelial function randomized, double-blind, placebo-controlled study. Nutr Metab Cardiovasc Dis. 2010 Nov;20(9):656-61. doi: 10.1016/j.numecd.2009.05.017. Epub 2009 Aug 20. PMID 19699071
- [Result] Faizi AK, Kornmo DW, Agewall S. Evaluation of endothelial function using finger plethysmography. Clin Physiol Funct Imaging. 2009 Sep;29(5):372-5. doi: 10.1111/j.1475-097X.2009.00882.x. Epub 2009 Jun 22. PMID 19552735
- [Result] Noa M, Mas R, Lariot C. Protective effect of policosanol on endothelium and intimal thickness induced by forceps in rabbits. J Med Food. 2007 Sep;10(3):452-9. doi: 10.1089/jmf.2006.232. PMID 17887938
- [Result] Moerland M, Kales AJ, Schrier L, van Dongen MG, Bradnock D, Burggraaf J. Evaluation of the EndoPAT as a Tool to Assess Endothelial Function. Int J Vasc Med. 2012;2012:904141. doi: 10.1155/2012/904141. Epub 2012 Feb 14. PMID 22500237
- [Result] Vizzardi E, Gavazzoni M, Della Pina P, Bonadei I, Regazzoni V, Sciatti E, Trichaki E, Raddino R, Metra M. Noninvasive assessment of endothelial function: the classic methods and the new peripheral arterial tonometry. J Investig Med. 2014 Aug;62(6):856-64. doi: 10.1097/JIM.0000000000000096. PMID 24945081
- [Result] Onkelinx S, Cornelissen V, Goetschalckx K, Thomaes T, Verhamme P, Vanhees L. Reproducibility of different methods to measure the endothelial function. Vasc Med. 2012 Apr;17(2):79-84. doi: 10.1177/1358863X12436708. Epub 2012 Mar 8. PMID 22402933